CLINICAL TRIAL: NCT02422836
Title: The Tolerability and Efficacy of a Three Product Anti-Aging Treatment Regimen in Subjects With Moderate to Severe Photodamage
Brief Title: Tolerability and Efficacy of Anti-Aging Treatment Regimen in Subjects With Photodamage
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US CosmeceuTechs, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Triple
Other Study IDs: USC-06-13.1
Record Dates: First submitted 2015-04-08; First posted 2015-04-21 (Estimated); Last update posted 2015-04-21 (Estimated); Status verified 2015-04

CONDITIONS: Skin Manifestations
Keywords: photodamage; fine lines; wrinkles; dyschromia
MeSH Terms: conditions — Skin Manifestations

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- Three Product Anti-Aging Regimen (Experimental): Three Product Anti-Aging Treatment Regimen:
  Cream Skin Cleanser RD04033B, twice daily, 8 weeks; Anti-aging Cream RD04034B, twice daily, 8 weeks; and Sunscreen SPF 50 RD04036, once daily, reapply as needed, 8 weeks
  Interventions: Other: Three Product Anti-Aging Treatment Regimen

INTERVENTIONS:
Other: Three Product Anti-Aging Treatment Regimen — Cream Skin Cleanser RD04033B, twice daily, 8 weeks; Anti-aging Cream RD04034B, twice daily, 8 weeks; and Sunscreen SPF 50 RD04036, once daily, reapply as needed, 8 weeks
  Other Names: Anti-aging Cream; Sunscreen SPF 50; Cream Skin Cleanser

SUMMARY:
The subjects will use the test skincare products. This is a full face, twice daily application study, with digital photos and expert grader evaluations at Baseline, 4 and 8 week periods. If the subject meets the study criteria and is enrolled, they will be instructed at screening visit to discontinue the use of any facial products (except dry mineral foundation and eye make-up) for seven (7) days before beginning the study (referred to as the "washout" period). They will return to the site for the baseline visit 2 after the required 7 day washout period (visit can occur within 1 week after screening visit).

DETAILED DESCRIPTION:
After the subjects properly consent to participation and are determined eligible, the study coordinator will review the subjects' medical history and obtain demographics. The Principal Investigator (PI) or designee (expert grader) will examine the subjects to determine their appropriateness for study inclusion.

At the Screening visit (Visit 1, Day -10 to -7), the subjects will be assessed by the PI or designee to confirm inclusion into the study. Expert grading and Canfield VISIA CR photographic documentation (all flash modes including RBX) will be performed at baseline (Visit 2, Day 0), Week 4 (Visit 3, Day 28 ± 7 days), and Week 8 (Visit 4, Day 56 ± 7 days).

Subjects who, in the PI's or designee's opinion, appear to be experiencing product related adverse reactions may be discontinued at any time during the study. The subjects' home care treatment products (the items included in the kit) will be performed at home, at the times and in the manner described in the instructions provided.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must be diagnosed by the investigator or expert grader to have moderate to severe lines/wrinkles (Grade 3 or higher, determined by the Glogau Scale).
2. Subjects must be 35 - 65 years of age with no known medical conditions that, in the investigator's opinion, may interfere with study participation.
3. Sexually active females of childbearing potential participating in the study must agree to use a medically-acceptable method of contraception while receiving study product. A woman of childbearing potential is defined as one who is biologically capable of becoming pregnant; including perimenopausal women who are less than 2 years from their last menses. Exception: Sexually inactive females of childbearing potential are not required to practice a reliable method of contraception and may be enrolled at the investigator's discretion, provided that they understand the possible risks involved in getting pregnant during the study and are counseled to remain sexually inactive for the duration of the study or to practice a reliable method of contraception if becoming sexually active during the study.
4. Subjects must sign a written informed consent.

Exclusion Criteria:

1. Any dermatologic disorder, which in the investigator's opinion, may interfere with the accurate evaluation of the subject's facial skin. Examples of such disorders include severe acne vulgaris, acne conglobata, acne fulminans, facial seborrheic dermatitis, and lupus erythematosus.
2. Subjects who have demonstrated a previous hypersensitivity reaction to any of the ingredients of the study products.
3. Concurrent therapy with any medication either topical or oral that might, in the investigator's opinion, interfere with the study.
4. Subjects who are not willing to discontinue their normal facial cosmetics during the study period. The subjects' dry mineral foundation and eye make-up are permitted, no liquid foundation; no other facial products other than the provided skincare products may be used.
5. Subjects who have used anti-aging skincare products (cosmetic and drug products with any of the following ingredients: AHA, Salicylic Acid, Vitamins A, Retin-A, Vitamin C, Growth Factors or Peptides, Antioxidants such as Idebenone, CoffeeBerry, CE Ferulic, Phloretin, etc.) within the last 3 months and during the course of the study.
6. Subjects with recent history in the past 6 months and during the course of the study of laser, chemical peels, microdermabrasion, or other medical treatments for the skin for anti-aging.
7. Subjects who are pregnant, breast feeding or planning a pregnancy during the study period.
8. Subjects who are unwilling or unable to comply with the requirements of the protocol.
9. No sun-bathing, use of sun lamps or tanning beds is permitted during the entire duration of the study.
10. Participation in another research study (currently or within the last 30 days).
11. All volunteers will sign the consent forms after being informed as to their obligations and risks that they might encounter as a participant in this study.

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2013-02; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Glogau Photodamage Scale: the change between the photodamage grade at Week 4 and Week 8 compared to the photodamage grade at the Baseline Visit. | 8 weeks
  The Glogau Photodamage Scale (Type I: No wrinkles, Type II: Wrinkles in motion, Type III: Wrinkles at rest, Type IV: Only wrinkles) represents a qualitative assessment to measure the severity of photodamage and wrinkles. Photodamage was graded at the Screening Visit (Day -10 to Day -7), Baseline Visit (Day 0), Week 4 Visit (Day 28), and Week 8 Visit (Day 56). The endpoint that was used to evaluate the primary objective of the study is the delta (change) between the photodamage grade at Week 4 Visit (Day 28) and Week 8 Visit (Day 56) compared to the photodamage grade at the Baseline Visit.

SECONDARY OUTCOMES:
Dryness and Flaking: the change between the dryness grade at Week 4 and Week 8 compared to the dryness grade at the Baseline Visit. | 8 weeks
  This parameter represents a visual assessment of skin dryness from normal skin (0/no dryness) to very severe dryness (5). Additionally, very marked visual flaking; very coarse scaling; cracking progressing to fissuring; marked thickening may be present.
Dyschromia: the change between the dyschromia grade at Week 4 and Week 8 compared to the dyschromia grade at the Baseline Visit. | 8 weeks
  This parameter represents a qualitative assessment of skin pigmentation from Normal (grade 0) to Severe (grade 5). Textural features likely to contribute to this grade include both red and brown patches of discoloration and other surface irregularities.
Stinging and Burning: the change between the stinging grade at Week 4 and Week 8 compared to the stinging grade at the Baseline Visit. | 8 weeks
  This parameter represents an assessment of any stinging or burning and relative duration of the sensation experienced by the subject when questioned by the Expert Grader. A scale of 0 to 5 as noted above can used to describe these findings when present.

CONTACTS AND LOCATIONS:
Overall Officials: Bruce Katz, MD, Principal Investigator — JUVA Skin & Laser Center / MediSpa

REFERENCES:
- [Derived] Katz BE, Lewis J, McHugh L, Pellegrino A, Popescu L. The Tolerability and Efficacy of a Three-product Anti-aging Treatment Regimen in Subjects with Moderate-to-severe Photodamage. J Clin Aesthet Dermatol. 2015 Oct;8(10):21-6. PMID 26557215